CLINICAL TRIAL: NCT01973127
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in Alcohol Dependent Patients: a Mechanistic Study.
Brief Title: Transcranial Magnetic Stimulation in the Treatment of Addiction
Acronym: MAGENTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IrisZorg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NISPA-IZ/MB22
Record Dates: First submitted 2013-10-22; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Alcohol Addiction
Keywords: alcohol; addiction; TMS; craving; use; rTMS; EEG; LPP; p300; ERN; SST; CCT; AAAT
MeSH Terms: conditions — Alcoholism; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum rTMS (Experimental): n=15. After detoxification of alcohol (maximum 4 days) rTMS treatment will start : 20 sessions (5 times during 4 weeks)of verum rTMS on the right dorsolateral prefrontal cortex.
  Measurements of all objectives at baseline and 2,4,8 and 12 weeks after start treatment.
  Interventions: Other: Verum rTMS
- Sham TMS (Sham Comparator): n=15. After detoxification of alcohol (maximum 4 days) rTMS treatment will start : 20 sessions (5 times during 4 weeks)of sham rTMS on the right dorsolateral prefrontal cortex.
  Measurements of all objectives at basleine and 2,4,8 and 12 weeks after start treatment.
  Interventions: Other: Sham rTMS

INTERVENTIONS:
Other: Verum rTMS — rTMS on the right dorsolateral prefrontal cortex. TMS procedure: The resting motor threshold (RMT) will be defined in each subject as the minimal stimulation intensity evoking an MEP of ≥ 0.05 mV in 50% of the trials in the muscle of the right thumb (M. abductor pollicis brevis). TMS will be conducted in the form of 'conventional rTMS', whereby 30 trains of 10 Hz pulses with a duration of 5 seconds and an inter-train interval of 25 seconds are applied to the righ dorsolateral prefrontal cortex (50 pulses per train, 6000 pulses per session). Used equipment: Magstim Rapid 2 device.
  Arms: Verum rTMS
Other: Sham rTMS — TMS procedure: The resting motor threshold (RMT) will be defined in each subject as the minimal stimulation intensity evoking an MEP of ≥ 0.05 mV in 50% of the trials in the muscle of the right thumb (M. abductor pollicis brevis). Like in verum TMS coil will be placed on the skull, but no magnetic field will be pulsed. Used equipment: Magstim Rapid 2 device.
  Arms: Sham TMS

SUMMARY:
The investigators hypothesize that repetitive transcranial magnetic stimulation (rTMS) on the right side of the head will make craving towards alcohol less severe in recently detoxified alcohol addicted patients.

Although there are successful treatment option to detoxify patients form their alcohol use, many patients tend to relapse. This relapse is mainly caused by a high level of (uncontrollable) craving towards alcohol. This aspect of addiction is with the existing options hard to treat, there is a great need of new successful treatment modalities. rTMS is a FDA approved treatment method for depression. Recently some small scale studies have shown promising results on rTMS in the treatment of addiction. In this study the investigators focus on alcohol addiction since it is the addiction with the highest morbidity and mortality in the Netherlands.

DETAILED DESCRIPTION:
In this study the investigators focus on three levels of interest: the biological level, the functional level and the clinical level. The investigators will measure the effect of rTMS directly on brain activity through EEG recording. The investigators investigate its effects on cognitive performance through the use of neuropsychological computer tasks. The investigators will address clinical behavior (craving and alcohol use) with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed males between 23-65 years of age
* A primary diagnose of alcohol dependence (meeting the DSM-IV-TR criteria 303.90/ICD-10 F10.2)
* Written consent for participation of the study.

Exclusion Criteria:

* MATE outcome <4 (as extracted from part 4 MATE at enrollment phase)MATE= Dutch screening instrument on (among others) addiction severity
* Presence of a current or past relevant somatic or neurological disorder
* Meeting the DSM-IV-TR criteria for a current bipolar disorder, schizophrenia, anxiety disorder or moderate to severe depressive disorder. These disorders would be a possible great confounder. Measured with the MINI-plus.
* Meeting the DSM-IV-TR criteria for current (in the past 2 weeks) dependence of substances other than alcohol, nicotine or caffeine. Information present in MATE.
* Participant-bound factors that may endanger participants or may jeopardize study adherence, because of failure to understand and/or comply with instructions (e.g. current, disruptive symptoms such as psychotic symptoms or severe cognitive impairment)
* Contra-indications resulting from the use of rTMS:

  * Epilepsy, convulsion or seizure
  * Serious head trauma or brain surgery
  * Large or ferromagnetic metal parts in the head (except for a dental wire)
  * Implanted cardiac pacemaker or neurostimulator

Ages: 23 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The change from baseline on the amplitude of the LPP at 8 weeks | 8 weeks after start of treatment.
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Late Positive Potentials (LPP) (P300 and Slow Potential (SP)) as measured with EEG at 8 weeks after start of treatment (baseline measurement).

SECONDARY OUTCOMES:
The change from baseline on the amplitude of the LPP at 2 weeks | 2 weeks after start of treatment
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Late Positive Potentials (LPP) (P300 and Slow Potential (SP)) as measured with EEG at 2 weeks after start of treatment (baseline measurement).
The change from baseline on the amplitude of the LPP at 4 weeks | 4 weeks after start of treatment
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Late Positive Potentials (LPP) (P300 and Slow Potential (SP)) as measured with EEG at 4 weeks after start of treatment (baseline measurement).
The change from baseline on the amplitude of the LPP at 12 weeks | 12 weeks after start of treatment
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Late Positive Potentials (LPP) (P300 and Slow Potential (SP)) as measured with EEG at 12 weeks after start of treatment (baseline measurement).
The change from baseline on the amplitude of the ERN at 2 weeks | 2 weeks after start of treatment
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Error Related Negativity (ERN) as measured with EEG at 2 weeks after start of treatment (baseline measurement).
The change from baseline on the amplitude of the ERN at 4 weeks | 4 weeks after start of treatment
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Error Related Negativity (ERN) as measured with EEG at 4 weeks after start of treatment (baseline measurement).
The change from baseline on the amplitude of the ERN at 8 weeks | 8 weeks after start of treatment
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Error Related Negativity (ERN) as measured with EEG at 8 weeks after start of treatment (baseline measurement).
The change from baseline on the amplitude of the ERN at 12 weeks | 12 weeks after start of treatment
  To investigate the effect of 20 sessions of rTMS on the change in amplitude of the Error Related Negativity (ERN) as measured with EEG at 12 weeks after start of treatment (baseline measurement).
Change from baseline on SST at 2 weeks | at 2 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 2 weeks follow-up, by conducting a Stop-Signal Task (SST)per computer.
Change from baseline on SST at 4 weeks | at 4 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 4 weeks follow-up, by conducting a Stop-Signal Task (SST)per computer.
Change from baseline on SST at 8 weeks | at 8 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 12 weeks follow-up, by conducting a Stop-Signal Task (SST) per computer.
Change from baseline on SST at 12 weeks | at 12 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 12 weeks follow-up, by conducting a Stop-Signal Task (SST) per computer.
Change from baseline on CCT at 2 weeks | at 2 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 2 weeks follow-up, by conducting a Columbia Card Task (CCT) per computer.
Change from baseline on CCT at 4 weeks | at 4 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 4 weeks follow-up, by conducting a Columbia Card Task (CCT) per computer.
Change from baseline on CCT at 8 weeks | at 8 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 8 weeks follow-up, by conducting a Columbia Card Task (CCT) per computer.
Change from baseline on CCT at 12 weeks | at 12 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 12 weeks follow-up, by conducting a Columbia Card Task (CCT) per computer.
Change from baseline on AAAT at 2 weeks | at 2 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 2 weeks follow-up, by conducting a Alcohol Approach Avoidance Task (AAAT) per computer.
Change from baseline on AAAT at 4 weeks | at 4 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 4 weeks follow-up, by conducting a Alcohol Approach Avoidance Task (AAAT) per computer.
Change from baseline on AAAT at 8 weeks | at 8 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 8 weeks follow-up, by conducting a Alcohol Approach Avoidance Task (AAAT) per computer.
Change from baseline on AAAT at 12 weeks | at 12 weeks after start treatement
  To investigate the effect of 20 sessions of rTMS on the change in cognitive performance at 12 weeks follow-up, by conducting a Alcohol Approach Avoidance Task (AAAT) per computer.
Change form baseline on craving at 2 weeks after start treatment | at 2 weeks after start treatment
  To investigate the change of 20 sessions of rTMS in perceived patient reported craving at 2 weeks after start treatment as measured with the Obsessive Compulsing Drinking Scale (OCDS), Alcohol Urge Questionnaire (AUQ) and a craving Visual Analogue Scale (VAS).
Change form baseline on craving at 4 weeks after start treatment | at 4 weeks after start treatment
  To investigate the change of 20 sessions of rTMS in perceived patient reported craving at 4 weeks after start treatment as measured with the Obsessive Compulsing Drinking Scale (OCDS), Alcohol Urge Questionnaire (AUQ) and a craving Visual Analogue Scale (VAS).
Change form baseline on craving at 8 weeks after start treatment | at 8 weeks after start treatment
  To investigate the change of 20 sessions of rTMS in perceived patient reported craving at 8 weeks after start treatment as measured with the Obsessive Compulsing Drinking Scale (OCDS), Alcohol Urge Questionnaire (AUQ) and a craving Visual Analogue Scale (VAS).
Change form baseline on craving at 12 weeks after start treatment | at 12 weeks after start treatment
  To investigate the change of 20 sessions of rTMS in perceived patient reported craving at 12 weeks after start treatment as measured with the Obsessive Compulsing Drinking Scale (OCDS), Alcohol Urge Questionnaire (AUQ) and a craving Visual Analogue Scale (VAS).
Change form baseline on alcohol use at 2 weeks after start treatment | at 2 weeks after start treatment
  To investigate the effect of 20 sessions of rTMS on the change in alcohol use 2 weeks from baseline by filling in a dairy on treatment days 5 times a week.
Change form baseline on alcohol use at 4 weeks after start treatment | at 4 weeks after start treatment
  To investigate the effect of 20 sessions of rTMS on the change in alcohol use 4 weeks from baseline by filling in a dairy on treatment days 5 times a week.
Change form baseline on alcohol use at 12 weeks after start treatment | at 8 weeks after start treatment
  To investigate the effect of 20 sessions of rTMS on the change in alcohol use 12 weeks from baseline by using the Alcohol Timeline Follow Back (TLFB) method.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Belgers, MD, Principal Investigator — IrisZorg
Locations (1):
- IrisZorg, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Feil J, Zangen A. Brain stimulation in the study and treatment of addiction. Neurosci Biobehav Rev. 2010 Mar;34(4):559-74. doi: 10.1016/j.neubiorev.2009.11.006. Epub 2009 Nov 13. PMID 19914283
- [Background] Barr MS, Farzan F, Wing VC, George TP, Fitzgerald PB, Daskalakis ZJ. Repetitive transcranial magnetic stimulation and drug addiction. Int Rev Psychiatry. 2011 Oct;23(5):454-66. doi: 10.3109/09540261.2011.618827. PMID 22200135
- [Background] Amiaz R, Levy D, Vainiger D, Grunhaus L, Zangen A. Repeated high-frequency transcranial magnetic stimulation over the dorsolateral prefrontal cortex reduces cigarette craving and consumption. Addiction. 2009 Apr;104(4):653-60. doi: 10.1111/j.1360-0443.2008.02448.x. Epub 2009 Jan 12. PMID 19183128
- [Derived] Belgers M, Markus W, Grasso F, Arns M, Van Eijndhoven P, Schellekens A. No Effects of rTMS on Performance Monitoring and Attentional Bias in Patients With Alcohol Use Disorder: A Pilot Study. Addict Biol. 2025 Nov;30(11):e70100. doi: 10.1111/adb.70100. PMID 41253702
- See also: site of addiction care organisation and sponsor — http://www.iriszorg.nl
- See also: site of university hospital where treatment takes place — http://www.umcn.nl
- See also: scientific institute related to the study — http://www.nispa.nl